CLINICAL TRIAL: NCT07298356
Title: Automated Applanation Tonometry - Updated
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106111_1
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma; Glaucoma, Suspect
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: In this 2 investigational methods (Fixed-force GAT and handheld tonometer) will be compared to the 2 standard methods (Standard GAT and pneumotonometer).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Standard GAT (Active Comparator): This is the gold-standard method for IOP measurement in clinical practice
  Interventions: Device: Standard GAT
- Fixed-force GAT (Experimental): From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a C-MOS camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter
  Interventions: Device: Fixed force GAT
- Upright applanating prototype (Experimental): With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter
  Interventions: Device: Upright applanating prototype
- Pneumotonometer (Active Comparator): This is another standard method for IOP measurement in clinical practice
  Interventions: Device: Pneumotonometer

INTERVENTIONS:
Device: Standard GAT — Standard Goldmann Applanation Tonometry (GAT): this is the standard method for IOP measurement in clinical practice
  Arms: Standard GAT
Device: Fixed force GAT — An investigational device similar to standard GAT
  Arms: Fixed-force GAT
Device: Upright applanating prototype — An investigational device, prism used in standard and fixed-force GAT is attached to a portable device
  Arms: Upright applanating prototype
Device: Pneumotonometer — This is a standard for checking eye pressure. A topical anesthetic (numbing agent). A probe will touch the front of the eye while the machine measures the eye pressure
  Arms: Pneumotonometer

SUMMARY:
Goldmann Applanation Tonometry (GAT) is considered the clinical gold standard for eye pressure measurements and yet it is known to be a subjective measurement with limited repeatability and limited portability. Another clinical standard for checking eye pressure is known as the pneumotonometer. This method is more objective but not portable. The purpose of this study is to develop new methods of measuring eye pressure that are more objective, reproducible and portable. In this study, we will be comparing the eye pressure measurements using 2 investigational methods to GAT and pneuumotonometer.

DETAILED DESCRIPTION:
This is a prospective study. Patients presenting for their scheduled eye appointments will be recruited by verbal communication. Following informed consent, intraocular pressure (IOP) measurements will be made by the following methods:

Standard Goldmann Applanation Tonometry (GAT): this is the standard method for IOP measurement in clinical practice. The eye is given topical fluorescein/anesthetic, the GAT prism contacts the eye while the observer looks through the slit lamp machine ocular using blue light illumination to visual the applanation mires. The GAT dial is adjusted until mire alignment is achieved and the IOP measurement is read off the GAT dial.

Pneumotonometer: This is what is done in routine eye care. You will receive a topical anesthetic (numbing agent). A probe will touch the front of the eye while the machine measures the eye pressure.

Fixed force GAT: From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a complementary metal oxide semiconductor (C-MOS) camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter. A similar method using an iPod touch camera has been previously published by this PI.

Upright applanating prototype: With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter.

The order of the above 4 measurements will be randomized.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Presenting for a routine eye exam
* ≥ 18 years of age
* Able and willing to give consent

Exclusion Criteria:

* History of corneal scarring
* Active infection of the eye
* Ocular surface trauma or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) as measured by standard GAT | Baseline
  this is the standard method for IOP measurement in clinical practice. The eye is given topical fluorescein/anesthetic, the GAT prism contacts the eye while the observer looks through the slit lamp machine ocular using blue light illumination to visual the applanation mires. The GAT dial is adjusted until mire alignment is achieved and the IOP measurement is read off the GAT dial.
Intraocular pressure (IOP) as measured by fixed force GAT | Baseline
  From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a C-MOS camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular.
Intraocular pressure as measured by upright applanating | Baseline
  With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter.
Intraocular pressure as measured by supine Pneumotonometer | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wen, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No Currently, there is no plan to share data with other researchers.